CLINICAL TRIAL: NCT06469203
Title: Oxytocin Effectiveness in First Trimester Dilatation and Curettage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Ashdod Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0127-23-AAA
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-06

CONDITIONS: Missed Abortion
Keywords: missed abortion; vaginal bleeding; dilation and curretage; pregnancy termination; oxytocin
MeSH Terms: conditions — Abortion, Missed; Uterine Hemorrhage; Dilatation, Pathologic | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Women undergoing dilation and curettage, who meet the eligibility criteria for the study, will be divided into two groups. They will receive the assigned medication at the beginning of the procedure, after cervical dilation but before using suction curettage.
  Group 1: Participants will receive 100 ml of saline alone. Group 2: Participants will receive an intravenous infusion of 8 units of oxytocin diluted in 100 ml of saline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomization will be done by hospitals pharmacy. A total of 160 patients will be included in the sample size resulting in a net total of 80 patients per group as described below. Patients who choose to withdraw from the study will still be analyzed as intention-to-treat patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive 100 ml of saline alone.
  Interventions: Drug: Sodium Chloride 0.9% Inj
- Oxytocin (Experimental): Participants will receive an intravenous infusion of 8 units of oxytocin diluted in 100 ml of saline.
  Interventions: Drug: Oxytocin; Drug: Sodium Chloride 0.9% Inj

INTERVENTIONS:
Drug: Oxytocin — Women undergoing dilation and curettage, who meet the eligibility criteria for the study, will be divided into two groups. They will receive the assigned medication at the beginning of the procedure, after cervical dilation but before using suction curettage.
  Group 1: Participants will receive 100 ml of saline alone. Group 2: Participants will receive an intravenous infusion of 8 units of oxytocin diluted in 100 ml of saline.
  Arms: Oxytocin
Drug: Sodium Chloride 0.9% Inj — Women undergoing dilation and curettage, who meet the eligibility criteria for the study, will be divided into two groups. They will receive the assigned medication at the beginning of the procedure, after cervical dilation but before using suction curettage.
  Group 1: Participants will receive 100 ml of saline alone. Group 2: Participants will receive an intravenous infusion of 8 units of oxytocin diluted in 100 ml of saline.

SUMMARY:
The aim of this study is to investigate the impact of oxytocin on perioperative blood loss during the D&C procedure, as well as to assess early and late complications associated with it's use.

DETAILED DESCRIPTION:
Study Design

This study is a prospective randomized placebo-controlled double-blind trial. Women undergoing dilation and curettage, who meet the eligibility criteria for the study, will be divided into two groups. They will receive the assigned medication at the beginning of the procedure, after cervical dilation but before using suction curettage.

Group 1: Participants will receive 100 ml of saline alone. Group 2: Participants will receive an intravenous infusion of 8 units of oxytocin diluted in 100 ml of saline.

The medication bags will be prepared by the Assuta Ashdod University Hospital Pharmacy, coded with serial numbers, and randomized using computerized software. Both the investigators and patients will remain unaware of the composition of the distension medium to ensure blinding.

A total of 160 patients will be included in the sample size resulting in a net total of 80 patients per group as described below. Patients who choose to withdraw from the study will still be analyzed as intention-to-treat patients.

Inclusion Criteria:

All patients admitted to the OBGYN Assuta Ashdod Hospital for elective surgical termination of pregnancy due to missed miscarriages in the first trimester, with gestational age range of 6.0 to 11.6 weeks.

Patients aged 18 years and older who are capable to provide informed consent.

Exclusion criteria

* individual intolerance to oxytocin
* mullerian anomalies
* Fibroid uterus
* thrombophilia or coagulation disorders
* cardiovascular disease

Primary outcome

Perioperative Blood Loss Assessment:

We will assess perioperative blood loss by:

* Measuring the content collected in the vacuum apparatus after the procedure.
* Recording hemoglobin and hematocrit levels prior to the procedure.
* Measuring hemoglobin and hematocrit levels immediately after the procedure.
* Monitoring hemoglobin and hematocrit levels two weeks post-procedure.

Secondary outcomes

-perioperative complications according to the Dindo-Clavien scale

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the OBGYN Assuta Ashdod Hospital for elective surgical termination of pregnancy due to missed miscarriages in the first trimester, with gestational age range of 6.0 to 11.6 weeks.

Patients aged 18 years and older who are capable to provide informed consent.

Exclusion Criteria:

* individual intolerance to oxytocin
* mullerian anomalies
* Fibroid uterus
* thrombophilia or coagulation disorders
* cardiovascular disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — including pregnant women
Enrollment: 160 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Perioperative Blood Loss Assessment | 14 days
  We will assess perioperative blood loss by:
  * Measuring the content collected in the vacuum apparatus after the procedure.
  * Recording hemoglobin and hematocrit levels prior to the procedure.
  * Measuring hemoglobin and hematocrit levels immediately after the procedure.
  * Monitoring hemoglobin and hematocrit levels two weeks post-procedure.

SECONDARY OUTCOMES:
perioperative complications according to the Dindo-Clavien scale | 30 days
  perioperative complications according to the Dindo-Clavien scale

IPD SHARING:
Plan to Share IPD: No